CLINICAL TRIAL: NCT01322633
Title: Long-Term Prospective Observational Study of the Risk of Cancer Among Pantoprazole Users
Brief Title: Risk of Cancer Among Pantoprazole Users
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 3001A1-100034; B1791018
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Results first posted 2014-02-20 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-01

CONDITIONS: Esophagitis
Keywords: Pantoprazole; proton pump inhibitor; gastric cancer; digestive system cancer; cancer
MeSH Terms: conditions — Esophagitis; Stomach Neoplasms; Digestive System Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pantoprazole: Patients who received treatment with pantoprazole tablets for at least 240 days within a 12-month period from 2000 through 2003.
  Interventions: Other: Does not apply
- Other proton pump inhibitors: Patients who received treatment with any other proton pump inhibitor for at least 240 days within a 12-month period from 1996 through 2003.
  Interventions: Other: Does not apply

INTERVENTIONS:
Other: Does not apply — This is a non-interventional study, therefore the intervention type / name do not apply.
  Groups: Pantoprazole
Other: Does not apply — This is a non-interventional study, therefore the intervention type / name do not apply.
  Groups: Other proton pump inhibitors

SUMMARY:
The primary objective is to assess whether the risk of gastric cancer is increased in pantoprazole users compared to users of other proton pump inhibitors.

DETAILED DESCRIPTION:
All subjects who met the inclusion criteria were included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have used pantoprazole or other proton pump inhibitors, enrollment in the health maintenance organization for at least 6 months, age 18 years or older.

Exclusion Criteria:

* Use of any proton pump inhibitor before study entry, any cancer diagnosis recorded in the medical history, diagnosis of Zollinger-Ellison Syndrome in medical history.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with long-term exposure to pantoprazole and other proton pump inhibitors enrolled in the Northern California Kaiser Permanente health maintenance organization.
Sampling Method: Non-Probability Sample
Enrollment: 61864 (Actual)
Dates: Start 2004-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3001A1-100034&StudyName=Risk%20of%20Cancer%20Among%20Pantoprazole%20Users%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Pantoprazole: Participants enrolled in Kaiser Permanente Northern California (KPNC) health maintenance organization who received treatment with pantoprazole (Protonix, pantoprazole sodium) tablets as per standard clinical practice for at least 240 days within a 12-month period during 4 years (from 2000 to 2003) before the start of study, were observed for up to 7.5 years.
- Other Proton Pump Inhibitors (PPI): Participants enrolled in KPNC health maintenance organization who received treatment with any PPI other than pantoprazole (any combination of omeprazole, lansoprazole, rabeprazole, or esomeprazole) as per standard clinical practice for at least 240 days within a 12-month period during 8 years (from 1996 to 2003) before the start of study, were observed for up to 7.5 years.
Period: Overall Study
Arm/Group | Pantoprazole | Other Proton Pump Inhibitors (PPI)
Started | 34178 | 27686
Completed | 34178 | 27686
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all participants who met the inclusion criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pantoprazole | Other Proton Pump Inhibitors (PPI) | Total
Number analyzed (Participants) | 34178 | 27686 | 61864
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59 [49 to 71] | 60 [50 to 71] | 60 [49 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19033 | 15611 | 34644
  Male | 15145 | 12075 | 27220

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Gastric Cancer
Description: Incidence rate was expressed as cases per 100,000 person-years with 95 percent (%) confidence intervals. Incidence rates were estimated from 1 year after the index date and were censored at the earliest of following events: diagnosis of gastric cancer, death, withdrawal from KPNC membership or end of the study, whichever occurred first for pantoprazole group. For other PPI group, data was also censored in case participants switched to pantoprazole group. Index date: the earliest date at which participant had achieved 240 days of study drug exposure within a 12 month time period before the study start date. Person-year was estimated by calculating all of the years that participants in a study were followed. Person-year calculations were adjusted for anticipated mortality based on United States (US) life tables.
Time Frame: 1 year after index date up to diagnosis of gastric cancer, death, withdrawal from KPNC membership, date when other PPI participants switched to pantoprazole or end of the study (up to Year 7.5)
Population: Analysis population included all participants who met the inclusion criteria.
Measure: Number (95% Confidence Interval); unit: incidence per 100000 person-years
Arm/Group | Pantoprazole | Other Proton Pump Inhibitors (PPI)
Number analyzed (Participants) | 34178 | 27686
incidence per 100000 person-years | 19.88 [14.26 to 26.96] | 23.73 [12.97 to 39.81]
Statistical Analysis 1: Comparison: Pantoprazole vs Other Proton Pump Inhibitors (PPI); Analysis was based on hazard ratio using Cox proportional hazard regression method adjusted for sex, age, cumulative PPI dose, total years of PPI treatment, diabetes, hepatitis C, hepatitis B and year of index date; Test type: Superiority or Other; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.24 to 1.93]

2. Secondary Outcome: Incidence Rate of Composite Gastrointestinal Cancers
Description: Incidence rate was expressed as cases per 100,000 person-years with 95 percent (%) confidence intervals. Incidence rates were estimated from 1 year after the index date and were censored at the earliest of following events: diagnosis of cancer of colon, pancreas, liver or small intestine, death, withdrawal from KPNC membership or end of the study, whichever occurred first for pantoprazole group. For other PPI group, data was also censored in case participants switched to pantoprazole group. Index date: the earliest date at which participant had achieved 240 days of study drug exposure within a 12 month time period before the study start date. Person-year was estimated by calculating all of the years that participants in a study were followed. Person-year calculations were adjusted for anticipated mortality based on United States (US) life tables.
Time Frame: 1 year after index date up to diagnosis of gastrointestinal cancer, death, withdrawal from KPNC membership, date when other PPI participants switched to pantoprazole or end of the study (up to Year 7.5)
Population: Analysis population included all participants who met the inclusion criteria.
Measure: Number (95% Confidence Interval); unit: incidence per 100000 person-years
Arm/Group | Pantoprazole | Other Proton Pump Inhibitors (PPI)
Number analyzed (Participants) | 34178 | 27686
incidence per 100000 person-years | 168.41 [151.13 to 187.12] | 129.25 [101.84 to 161.78]
Statistical Analysis 1: Comparison: Pantoprazole vs Other Proton Pump Inhibitors (PPI); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.65 to 1.40]

3. Secondary Outcome: Incidence Rate of Overall Cancer
Description: Incidence rate was expressed as cases per 100,000 person-years with 95 percent (%) confidence intervals. Incidence rates were estimated from 1 year after the index date and were censored at the earliest of following events: diagnosis of any type of cancer (excluding non-melanoma skin cancers), death, withdrawal from KPNC membership or end of the study, whichever occurred first for pantoprazole group. For other PPI group, data was also censored in case participants switched to pantoprazole group. Index date: the earliest date at which participant had achieved 240 days of study drug exposure within a 12 month time period before the study start date. Person-year was estimated by calculating all of the years that participants in a study were followed. Person-year calculations were adjusted for anticipated mortality based on United States (US) life tables.
Time Frame: 1 year after index date up to diagnosis of any cancer, death, withdrawal from KPNC membership, date when other PPI participants switched to pantoprazole or end of the study (up to Year 7.5)
Population: Analysis population included all participants who met the inclusion criteria.
Measure: Number (95% Confidence Interval); unit: incidence per 100000 person-years
Arm/Group | Pantoprazole | Other Proton Pump Inhibitors (PPI)
Number analyzed (Participants) | 34178 | 27686
incidence per 100000 person-years | 1465.21 [1412.12 to 1519.79] | 1369.88 [1275.12 to 1469.82]
Statistical Analysis 1: Comparison: Pantoprazole vs Other Proton Pump Inhibitors (PPI); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.93 to 1.21]

ADVERSE EVENTS:
Description: The study used de-identified patient-level electronic health related databases (e-HRD), in which it was not possible to link a particular product and medical event for any participant. Thus, minimum criteria for reporting an adverse event were not available and adverse events were not reportable as individual AE reports.
Arm/Group | Pantoprazole | Other Proton Pump Inhibitors (PPI)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.